CLINICAL TRIAL: NCT02402829
Title: A Study Comparing Factor Level and Inhibitor Titer Testing Results Drawn From Central Venous Lines and Venipuncture
Acronym: CVL#2
Status: Terminated | Type: Observational
Why Stopped: lack of participation or interest in other sites.
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Other Study IDs: 14040182
Record Dates: First submitted 2015-01-30; First posted 2015-03-30 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Hemophilia A; Factor VIII Deficiency; Hemophilia; Hemophilia B; Factor IX Deficiency
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemophilia Patients: Subjects diagnosed with moderate or severe Hemophilia A or B who use a central venous line (CVL) for regular prophylaxis factor infusions and are at the clinic for a standard of care visit. As part of the study all subjects will have blood drawn through their CVL and will also undergo a peripheral vein blood draw.
  Interventions: Procedure: Peripheral Vein Blood draw

INTERVENTIONS:
Procedure: Peripheral Vein Blood draw — Drawing blood through a peripheral vein in the arm.

SUMMARY:
The purpose of this research study is to see if factor levels and inhibitor levels in Hemophilia A and B subjects are accurate when they are drawn from a central venous line (CVL) instead of from a peripheral stick.

DETAILED DESCRIPTION:
Patients with hemophilia A and B sometimes require the placement of a central venous line (CVL). A CVL is a medical device that is placed into a vein that gives easier access to a vein either for a blood draw or to give factor replacement product.

Patients with hemophilia are usually seen by the hemophilia doctor every year at the annual comprehensive clinic visit. As part of this visit, the doctor usually orders routine blood tests, including the factor level and inhibitor titer.The factor level and inhibitor blood tests are always taken through a "peripheral stick." A peripheral stick means that a small needle is inserted into a vein in order to obtain a blood sample. The CVL is not used for these blood draws. This is because the investigators don't know if the infusion of factor replacement product and heparin (a blood thinning drug used to flush the line after a factor infusion) can cause the blood sample results to be incorrect. The current practice is to take blood through a needle stick in the vein because the investigators can be sure that the results are accurate.

When blood draws are taken through a peripheral stick, it can cause children with hemophilia to be very anxious because of the pain involved with a needle stick. Also, the needle stick can sometimes cause a bleed, which may require treatment.

The purpose of this research study is to see if factor levels and inhibitor levels are accurate when they are drawn from a CVL instead of from a peripheral stick.

ELIGIBILITY:
Inclusion Criteria:

* Children and adults with hemophilia A or B, ages 1-21 who have CVLs for factor infusion and who are prescribed factor prophylaxis for treatment of their bleeding disorder will be included.
* Subjects will be recruited from active patients at federally funded hemophilia treatment centers (HTCs).

Exclusion Criteria:

* None

Ages: 1 Year to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects with moderate or severe Hemophilia A or B.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2014-11; Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Evaluate the equivalence between coagulation labs drawn from central venous line to those drawn peripherally. Primary measurements will be done on factor levels resulted as percent of normal, and inhibitor titers resulted in Bethesda Units (BU). | within 15 minutes pre-infusion of a factor replacement product
Evaluate the equivalence between coagulation labs drawn from central venous line to those drawn peripherally. Primary measurements will be done on factor levels resulted as percent of normal, and inhibitor titers resulted in Bethesda Units (BU). | 15 minutes after the infustion of a factor replacement product

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States